CLINICAL TRIAL: NCT04296643
Title: Medical Masks Versus N95 Respirators to Prevent 2019 Novel Coronavirus Disease (COVID-19) in Healthcare Workers: A Randomized Trial
Brief Title: Medical Masks vs N95 Respirators for COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20006014
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus; N95; Medical Mask
MeSH Terms: conditions — Coronavirus Infections | interventions — N95 Respirators

STUDY DESIGN:
Intervention Model Description: pragmatic, randomized, open-label, multicentre, noninferiority trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and laboratory assessors were blinded to the group assignment, but it was not possible to conceal the identity of the medical mask or N95 respirator assignment to the study staff or participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Mask (Experimental): Medical Mask worn when providing care to patient with febrile respiratory illness
  Interventions: Device: Medical Mask
- N95 respirator (Active Comparator): N95 respirator worn when providing care to patient with febrile respiratory illness
  Interventions: Device: N95 respirator

INTERVENTIONS:
Device: Medical Mask — Medical Mask (known also as Surgical Mask)
  Arms: Medical Mask
Device: N95 respirator — N95 respirator
  Arms: N95 respirator

SUMMARY:
A randomized controlled trial in which health care workers will be randomized to either medical masks or N95 respirators when providing care to patients with COVID-19.

DETAILED DESCRIPTION:
A randomized controlled trial in which health care workers will be randomized to either medical masks or N95 respirators when providing medical care to patients with COVID-19. This multi-centre randomized controlled trial will assess whether medical masks are non-inferior to N95 respirators when health care workers provide care involving non-aerosol generating procedures. Health care workers will be randomized to either use of a medical mask or to a fit-tested N95 respirator when providing care for patients with febrile respiratory illness. Health care workers randomly assigned to the N95 respirator group will be instructed to use a fit-tested National Institute for Occupational Safety and Health-approved N95 respirator when providing routine care to patients with COVID-19 or suspected COVID-19. Participants will use the type of device they were allocated to, either a medical mask or an N95 respirator, for 10 weeks, however, health care workers can also use the N95 respirator at any time based on a point-of-care risk assessment. Universal masking is the policy implemented at each study site. Extended and re-use of N95 respirators will be permitted if the local situation requires it. The primary outcome is laboratory confirmed RT-PCR COVID-19 among participants.

A nasopharyngeal swab will be obtained if any one of the following symptoms or signs is present: fever (≥38 C), cough, or shortness of breath, or if 2 of the following are present: fatigue, myalgia, headache, dizziness, expectoration, sore throat, diarrhea, nausea, vomiting, abdominal pain, runny nose, altered taste or smell, conjunctivitis, or painful swallowing.

Participants that receive a COVID-19 vaccine after enrollment with efficacy of > 50% for the circulating strain will continue to be followed until 2 weeks after the first dose of the vaccine. All other participants will be followed for 10 weeks.

Self-reporting of hand hygiene and the use of external monitors, where feasible, will be used to collect basic hand hygiene data.

The sample size is 1,010 participants. This will allow 90% power at an alpha (one sided) of 0.05 and to account for participants who may not have completed 10 weeks because of COVID-19 mRNA vaccination.

Changes made to the protocol prior to May 4, 2020, which was prior to the start of enrollment:

* Eligibility criteria expanded from nurses who provide direct patient care to health care workers that provide direct patient care.
* Allowed extended and re-use of N95 respirators if the local situation required it.
* Added self-reporting of hand hygiene and the use of external monitors if feasible.
* Reduced the duration of follow up from 12 weeks to 10 weeks

Changes made on or after May 4, 2020:

* Expanded the criteria for the requirement of swabs to detect COVID-19 by adding runny nose, altered taste or smell, and conjunctivitis and also asked for a swab for fever, cough, or shortness of breath alone OR for two of the previously listed symptoms or signs (May 19, 2020).
* Added previously known COVID infection as an exclusion (October, 30, 2020).
* Added receipt of a COVID-19 vaccine with efficacy of > 50% as an exclusion (October 30, 2020).
* Allowed those participants that received a COVID-19 vaccine after enrollment with efficacy of > 50% for the circulating strain to continue to be followed until 2 weeks after the first dose of the vaccine (December 17, 2020).
* Increased the sample size to 1,010 participants to allow 90% power at an alpha (one sided) of 0.05 and to account for participants who may not have completed 10 weeks because of COVID-19 mRNA vaccination (July 26, 2021).
* Added wording to capture implementation since May 4th, 2020, "Where the policy of the healthcare setting has been universal use of a facemask, that is wearing a facemask at all times when in the hospital, then the facemask participants were randomized to will be used." (December 27, 2021)

ELIGIBILITY:
Inclusion Criteria:

* Health care workers who provide direct care to patients with suspected or confirmed COVID-19 in specialized COVID-19 units and in emergency departments, medical units, pediatric units, and long-term care facilities
* Health care workers are required to spend 60% or more of their time doing clinical work when enrolled.

Exclusion Criteria:

* Unable to pass or do not have a valid fit test within the past 24 months
* One or more high-risk comorbidities for COVID-19 (hypertension, cardiac disease, pulmonary disease, chronic kidney disease, diabetes, chronic liver disease, actively treated cancer, or immunosuppression due to illness or medications)
* Previous laboratory confirmed clinical diagnosis of COVID-19 at the time of
* Received 1 or more doses of a COVID-19 vaccine with greater than 50% efficacy for the circulating strain (for example, mRNA or vector-based COVID-19 vaccine against the original SARS-CoV-2 strain).
* working in intensive care units.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1009 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
RT-PCR confirmed COVID-19 infection | 10 weeks
  Number of participants with RT-PCR confirmed COVID-19 infection

SECONDARY OUTCOMES:
Acute respiratory illness | 10 weeks
  Number of participants with acute respiratory illness
Absenteeism | 10 weeks
  Number of participants with absenteeism
Lower respiratory infection | 10 weeks
  Number of participants with lower respiratory infection
Pneumonia | 10 weeks
  Number of participants with pneumonia
ICU admission | 10 weeks
  Number of participants with ICU admission
Mechanical ventilation | 10 weeks
  Number of participants needing mechanical ventilation
Death | 10 weeks
  Number of participants that died

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Loeb, Principal Investigator — McMaster University
Locations (15):
- Canada (12):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Brantford General Hospital, Brantford, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Hopital Montfort, Ottawa, Ontario
  - Niagara Health Services, Saint Catherines, Ontario
  - St. Joe's Unity Health, Toronto, Ontario
  - St. Mike's Unity Health, Toronto, Ontario
  - Montreal University Health Centre, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
- Fayoum General Hospital, Al Fayyum, Egypt
- Golden Care LTCF, Tzrifin, Israel
- Dr. Ziauddin Hospital, Karachi, Pakistan

REFERENCES:
- [Derived] Loeb M, Bartholomew A, Hashmi M, Tarhuni W, Hassany M, Youngster I, Somayaji R, Larios O, Kim J, Missaghi B, Vayalumkal JV, Mertz D, Chagla Z, Cividino M, Ali K, Mansour S, Castellucci LA, Frenette C, Parkes L, Downing M, Muller M, Glavin V, Newton J, Hookoom R, Leis JA, Kinross J, Smith S, Borhan S, Singh P, Pullenayegum E, Conly J. Medical Masks Versus N95 Respirators for Preventing COVID-19 Among Health Care Workers : A Randomized Trial. Ann Intern Med. 2022 Dec;175(12):1629-1638. doi: 10.7326/M22-1966. Epub 2022 Nov 29. PMID 36442064
- [Derived] Schunemann HJ, Akl EA, Chou R, Chu DK, Loeb M, Lotfi T, Mustafa RA, Neumann I, Saxinger L, Sultan S, Mertz D. Use of facemasks during the COVID-19 pandemic. Lancet Respir Med. 2020 Oct;8(10):954-955. doi: 10.1016/S2213-2600(20)30352-0. Epub 2020 Aug 3. No abstract available. PMID 32758441